CLINICAL TRIAL: NCT04095039
Title: HiLo: Pragmatic Trial of Higher vs Lower Serum Phosphate Targets in Patients Undergoing Hemodialysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility of enrollment and futility of separation between study arms
Sponsor: Duke University (Other)
Collaborators: Northwestern University (Other); University of Pennsylvania (Other); Davita Clinical Research (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Association of Kidney Patients (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100325; 5UH3DK118748-05 (NIH)
Record Dates: First submitted 2019-09-10; First posted 2019-09-19 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2023-07

CONDITIONS: All-cause Mortality; Hospitalization
Keywords: All-cause Mortality; All-cause hospitalization; Phosphate management; Hemodialysis
MeSH Terms: interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hi Arm (Experimental): Patients to allow blood serum phosphate levels to rise to 6.5 mg/dl or above
  Interventions: Procedure: Hemodialysis
- Lo Arm (No Intervention): Patients to titrate blood serum phosphate levels to the standard <5.5mg/dl

INTERVENTIONS:
Procedure: Hemodialysis — Patients in both arms will undergo hemodialysis to remove phosphate from the blood; however, patients in the Hi Arm will only be titrated down to no lower than 6.5mg/dl
  Arms: Hi Arm

SUMMARY:
HiLo will be a pragmatic, open-label, multicenter, clinical trial with individual level randomization of ~4400 patients with ESRD undergoing in-center maintenance hemodialysis at 120-150 units maintained by two dialysis organizations that care for a substantial proportion of the US dialysis population. The 1st objective of HiLo is to test the following primary and secondary hypotheses of HiLo:

Primary hypothesis: Compared to the current standard approach of targeting serum phosphate levels of <5.5 mg/dl, less stringent control of serum phosphate to target levels of ≥6.5 mg/dl will yield a reduction in the hierarchical composite outcome of time to all-cause mortality and all-cause hospitalization among patients with ESRD undergoing hemodialysis.

Secondary hypothesis: The main secondary hypotheses are that less stringent control of serum phosphate will reduce risk of all-cause mortality as well as the risk of all-cause hospitalization (individually) compared to the current standard approach of strict phosphate control (superiority analysis). In addition, the trial will test the secondary hypotheses that less stringent control of serum phosphate will result in increased serum albumin and protein catabolic rate (PCR), as markers of diet and nutrition.

The 2nd objective of HiLo is to conduct a second-generation pragmatic clinical trial in dialysis. In partnership with two dialysis provider organizations, demonstrate the following for a trial embedded in clinical care delivery:

1. Feasibility of obtaining informed consent using electronic devices (e-consent)
2. Use of a single IRB of record for hundreds of dialysis facilities
3. Successful implementation of a trial-driven treatment algorithm by dietitians at the participating dialysis units
4. Harmonization of data from a large for-profit dialysis provider and an academically-owned small dialysis provider
5. Effective monitoring of trial implementation using a centralized approach

DETAILED DESCRIPTION:
Pragmatic Trial Demonstration Goals

The HiLo Trial is one of the pragmatic trial demonstration projects of the NIH Health Care Systems (HCS) Research Collaboratory. These demonstration projects are intended to be large clinical trials that are conducted within the clinical care environment and evaluate interventions implemented by care providers and relying as much as possible on data obtained as part of routine clinical care. HiLo has the following demonstration project goals:

1. To implement an electronic consent process;
2. To use a single IRB of record to oversee hundreds of dialysis facilities;
3. To implement a trial-driven treatment algorithm by dietitians at the participating dialysis units
4. To harmonize across 2 different dialysis providers data elements obtained though clinical care;
5. To monitor safety without using individual adverse event reporting.

HiLo will individually randomize participants using facility-level stratification to achieve balance across the two arms. Stratification will be 1:1 within each facility.

Participants will be followed for up to 27 (enter at enrollment end) - 45 (enter at enrollment start) months.

Two phosphate titration protocols will be used that have the same "look and feel" as those used in practice in an effort to sustain a mean time-averaged difference in serum phosphate between the two arms of ≥1 mg/dl:

1. Low serum phosphate target that is consistent with current standard of care: The goal is to titrate and maintain serum phosphate to <5.5 mg/dl.
2. Higher serum phosphate target that is the intervention strategy: The goal is to titrate and maintain serum phosphate to ≥6.5 mg/dl by setting a serum phosphate threshold >7.0 mg/dl when binders will be initiated, as has been done previously.

A mean serum phosphate of 4.8-5.2 is anticipated in the low arm and 6.5-6.8 in the high arm, as observed in two pilot clinical trials.Since serum phosphate is 4-7 mg/dl in most patients with ESRD, ≥1 mg/dl difference equates with a ≥33% difference within the modifiable range of time-averaged phosphate exposure. Specific binder choices will be relegated to the discretion of local providers based on local practice.

Planned Enrollment and randomization Enrollment of the first subject - 03/13/2020 (Actual) 25% of planned enrollment recruited - 06/30/2022 (Anticipated) 50% of planned enrollment recruited - 10/30/2022 (Anticipated) 75% of planned enrollment recruited - 03/31/2023 (Anticipated) 100% of planned enrollment recruited - 09/30/2023 (Anticipated) 6.4. Completion of primary endpoint data analyses - 11/30/2024 (Anticipated) 6.5. Reporting of results in ClinicalTrials.gov - 1/31/2025 (Anticipated)

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Undergoing 3 times weekly in-center hemodialysis and have been receiving dialysis treatment for at least 3 months
* Able to provide written informed consent

Exclusion Criteria:

* Pregnancy
* In-center Nocturnal
* Calciphylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myles Wolf, MD, MMSc, Principal Investigator — Duke Nephrology
Locations (84):
- United States (84):
  - DaVita Ensley, Birmingham, Alabama
  - DaVita Phoenix Dialysis, Phoenix, Arizona
  - DaVita Ouachita Valley, Camden, Arkansas
  - DaVita South Arkansas, El Dorado, Arkansas
  - DaVita Fayetteville, Fayetteville, Arkansas
  - DaVita Mena, Mena, Arkansas
  - DaVita Springdale, Springdale, Arkansas
  - DaVita El Dorado Dialysis, Long Beach, California
  - DaVita San Diego South, San Diego, California
  - DaVita Hamden, Hamden, Connecticut
  - DaVita Middlesex, Middletown, Connecticut
  - DaVita New Britain, New Britain, Connecticut
  - DaVita Torrington, Torrington, Connecticut
  - DaVita Celebration Dialysis, Kissimmee, Florida
  - DaVita Troup County Dialysis, La Grange, Georgia
  - DaVita Thomaston Dialysis, Thomaston, Georgia
  - DaVita Stony Island, Chicago, Illinois
  - DaVita West Joliet, Joliet, Illinois
  - DaVita Vincennes Dialysis, Vincennes, Indiana
  - DaVita Northeast Cambridge, Cambridge, Massachusetts
  - DaVita Wellington Circle, Medford, Massachusetts
  - DaVita Highland Park, Highland Park, Michigan
  - DaVita Arden Hills, Arden Hills, Minnesota
  - DaVita Bloomington, Bloomington, Minnesota
  - DaVita Burnsville, Burnsville, Minnesota
  - DaVita Cass Lake, Cass Lake, Minnesota
  - DaVita Coon Rapids, Coon Rapids, Minnesota
  - DaVita Cottage Grove, Cottage Grove, Minnesota
  - DaVita Moorehead, Dilworth, Minnesota
  - DaVita Eden Prairie, Eden Prairie, Minnesota
  - DaVita Faribault, Faribault, Minnesota
  - DaVita East River Road, Fridley, Minnesota
  - DaVita Glencoe, Glencoe, Minnesota
  - DaVita Historical Hastings, Hastings, Minnesota
  - DaVita Lakeville, Lakeville, Minnesota
  - DaVita Maple Grove, Maple Grove, Minnesota
  - DaVita Minneapolis Uptown, Minneapolis, Minnesota
  - DaVita Minnetonka, Minnetonka, Minnesota
  - DaVita New Ulm, New Ulm, Minnesota
  - DaVita Northfield, Northfield, Minnesota
  - DaVita Redwood Falls, Redwood Falls, Minnesota
  - DaVita Richfield, Richfield, Minnesota
  - DaVita Rochester, Rochester, Minnesota
  - DaVita St. Louis Park, Saint Louis Park, Minnesota
  - DaVita St. Paul, Saint Paul, Minnesota
  - DaVita Sun Ray, Saint Paul, Minnesota
  - DaVita University Riverside, Saint Paul, Minnesota
  - DaVita Scott County, Savage, Minnesota
  - DaVita West St. Paul, West Saint Paul, Minnesota
  - DaVita Wyoming, Wyoming, Minnesota
  - DaVita Omaha West Dialysis, Omaha, Nebraska
  - DaVita Centennial, Las Vegas, Nevada
  - DaVita Pahrump, Pahrump, Nevada
  - DaVita Bronx, The Bronx, New York
  - DaVita Orchard Park Dialysis, West Seneca, New York
  - Burlington Dialysis, Burlington, North Carolina
  - North Burlington Dialysis, Burlington, North Carolina
  - Durham Dialysis, Durham, North Carolina
  - Bull City Dialysis, Durham, North Carolina
  - Durham West Dialysis, Durham, North Carolina
  - Southpoint Dialysis, Durham, North Carolina
  - DaVita Goldsboro South Dialysis, Goldsboro, North Carolina
  - Vance County Dialysis, Henderson, North Carolina
  - Kerr Lake, Louisburg, North Carolina
  - DaVita Reidsville Dialysis, Reidsville, North Carolina
  - DaVita Roxboro Dialysis, Roxboro, North Carolina
  - DaVita Southern Pines Dialysis, Southern Pines, North Carolina
  - DaVita Fargo, Fargo, North Dakota
  - DaVita Midwest Fairborn, Fairborn, Ohio
  - DaVita Moore, Moore, Oklahoma
  - DaVita Tahlequah, Tahlequah, Oklahoma
  - DaVita McKeesport West, McKeesport, Pennsylvania
  - DaVita Radnor, Radnor, Pennsylvania
  - DaVita Blount Dialysis, Maryville, Tennessee
  - Renal Center of Waterton, Tyler, Texas
  - American Fork Dialysis, American Fork, Utah
  - DaVita Bountiful Dialysis, Bountiful, Utah
  - DaVita Farmington Bay Dialysis, Layton, Utah
  - Payson Dialysis, Payson, Utah
  - Provo Dialysis, Provo, Utah
  - DaVita Kolff, Salt Lake City, Utah
  - DaVita Sandy Dialysis, Sandy City, Utah
  - Sandy Dialysis, Taylorsville, Utah
  - DaVita Federal Way Dialysis, Federal Way, Washington

IPD SHARING:
Plan to Share IPD: Yes
Will share data in accordance with the NIH data sharing guidelines
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The Study Protocol SAP will be presented in a methods paper which is planned to be submitted to statistical professionals journals in the coming months. The CSR and the deidentified clinical database will be provided to the NIDDK data repository w/in 3 months of database lock.
Access Criteria: Access criteria will be maintained by the NIDDK.
URL: https://repository.niddk.nih.gov/home

REFERENCES:
- [Derived] Edmonston D, Isakova T, Dember LM, Waymyers S, Andersen D, Chan KE, Chakraborty H, Wolf M. Higher versus Lower Phosphate Targets for Patients Undergoing In-Center Hemodialysis: A Randomized Controlled Trial. J Am Soc Nephrol. 2025 Dec 1;36(12):2445-2455. doi: 10.1681/ASN.0000000765. Epub 2025 Jul 10. PMID 40638247
- [Derived] Fajol A, Faul C. The Pathologic Actions of Phosphate in CKD. Kidney360. 2025 Apr 17;6(6):1040-1049. doi: 10.34067/KID.0000000820. PMID 40241437
- [Derived] Edmonston DL, Isakova T, Dember LM, Brunelli S, Young A, Brosch R, Beddhu S, Chakraborty H, Wolf M. Design and Rationale of HiLo: A Pragmatic, Randomized Trial of Phosphate Management for Patients Receiving Maintenance Hemodialysis. Am J Kidney Dis. 2021 Jun;77(6):920-930.e1. doi: 10.1053/j.ajkd.2020.10.008. Epub 2020 Dec 3. PMID 33279558

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lo Arm | Hi Arm
Started | 441 | 352
Completed | 368 (Since Death is part of the primary endpoint, participants who died are considered to have completed the study) | 261 (Since Death is part of the primary endpoint, participants who died are considered to have completed the study)
Not Completed | 73 | 91
Not completed — Withdrawal by Subject | 2 | 16
Not completed — Transplanted | 21 | 24
Not completed — Transferred to Non-study Facility | 47 | 44
Not completed — Withdrawal from internvention target | 0 | 2
Not completed — Switch to peritoneal dialysis or home hemodialysis | 2 | 4
Not completed — Cacliphylaxis | 0 | 1
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lo Arm | Hi Arm | Total
Number analyzed (Participants) | 441 | 352 | 793
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (14.29) | 59.2 (15.00) | 60.3 (14.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 152 | 329
  Male | 264 | 200 | 464
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 45 | 92
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 382 | 295 | 677
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 19 | 34
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 4 | 6 | 10
  Black or African American | 181 | 146 | 327
  White | 180 | 129 | 309
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 58 | 48 | 106
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 441 | 352 | 793
PCR [Mean (Standard Deviation); unit: g/kg/day] | 1.0 (0.29) | 1.1 (0.32) | 1.1 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Hierarchical Composite Mortality and All Cause Hospitalization
Description: Hierarchical composite of time to all-cause mortality and all-cause hospitalization rate (total counts per person-years of follow-up) for the individually randomized cohort
Time Frame: up to 27 (enter at enrollment end) - 45 (enter at enrollment start) months
Population: Based on DSMB concerns we adjusted the randomization scheme from cluster-randomized to individual randomization due to concerns of self-selection. At the time that the trial was terminated, only 249 participants were individually randomized so we restricted our analysis to that population.
Measure: Number; unit: total number of events
Arm/Group | Lo Arm | Hi Arm
Number analyzed (Participants) | 125 | 124
total number of events
  All-cause mortality | 2 | 5
  All-cause Hospitalizations | 98 | 128
Statistical Analysis 1: Comparison: Lo Arm vs Hi Arm; Primary outcome is for the individually randomized cohort since DSMB had concerns about selection bias for the cluster-randomized population due to differences in baseline characteristics that leaned towards the arm objectives; Test type: Superiority; p = 0.077, Finkelstein-Schoenfeld method — p-value is based on a sample that is less than 10% of the planned sample size (planned n=4,000)

2. Secondary Outcome: Time to All-cause-mortality
Description: Time to all-cause-mortality from baseline for both cluster-randomized and individually randomized cohorts.
Time Frame: up to 27 (enter at enrollment end) - 45 (enter at enrollment start) months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Lo Arm | Hi Arm
Number analyzed (Participants) | 96 | 57
Years | 1.2 (0.72) | 1.4 (0.80)

3. Secondary Outcome: Hospitalization Days
Description: Total days hospitalized (Data reflects participants with valid, non-missing hospitalization start and end dates.)
Time Frame: up to 27 (enter at enrollment end) - 45 (enter at enrollment start) months
Population: Total days hospitalized from baseline for both cluster-randomized and individually randomized cohorts. (Data reflects participants with valid, non-missing hospitalization start and end dates)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lo Arm | Hi Arm
Number analyzed (Participants) | 441 | 352
Days | 27.9 (29.4) | 35.4 (46.1)

4. Secondary Outcome: Serum Albumin
Description: serum albumin as markers of diet and nutrition.
Time Frame: Baseline (days -30 - 0)
Population: Serum albumin at baseline for both cluster-randomized and individually randomized cohorts as a marker of diet and nutrition
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lo Arm | Hi Arm
Number analyzed (Participants) | 441 | 352
g/dL | 4.1 (0.35) | 4.1 (0.35)

5. Secondary Outcome: Protein Catabolic Rate (PCR)
Description: protein catabolic rate (PCR) as markers of diet and nutrition (g/kg/day).
Time Frame: Baseline (days -30 - 0)
Population: Protein catabolic rate at baseline for both cluster-randomized and individually randomized cohorts as a marker of diet and nutrition
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Hi Arm | Lo Arm
Number analyzed (Participants) | 441 | 352
g/kg/day | 1.0 (0.29) | 1.1 (0.32)

ADVERSE EVENTS:
Time Frame: All cause mortality was collected up to 45 months (27 months if the participant entered the study at enrollment end; up to 45 months if the participant entered at enrollment start). Additional adverse events were not collected.
Description: Among patients undergoing hemodialysis, adverse events of moderate or higher severity are extremely common and usually result in hospitalization (or death). Based on this information, and given that hospitalization is the primary outcome of HiLo, additional information on adverse events will not be collected.
Arm/Group | Lo Arm | Hi Arm
All-Cause Mortality (participants affected / at risk) | 94/316 | 52/228
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Trial was early terminated leading to less than 10% of the planned sample size being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT04095039/Prot_001.pdf
  • Statistical Analysis Plan (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT04095039/SAP_003.pdf
  • Informed Consent Form (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04095039/ICF_002.pdf